CLINICAL TRIAL: NCT03610750
Title: PRIDE SSA - Partnerships in Research to Implement and Disseminate Sustainable and Scalable Evidence Based Practices in Sub-Saharan Africa
Brief Title: Training Providers to Conduct PRIDES-sSA
Acronym: PRIDE-sSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Milton L. Wainberg, MD, Professor of Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 7485
Record Dates: First submitted 2018-03-13; First posted 2018-08-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Common Mental Disorders; Severe Mental Disorder
Keywords: Community Mental Health Care; Task-shifting
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Effectiveness-Implementation Hybrid 1 Trial
Who Masked: Investigator
Masking Description: De-identified aggregate clinic will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Specialty Care (Active Comparator): Psychiatric medications and evidence-based psychotherapies to be provided at a specialty mental clinic facilitated by psychiatric technicians, the mental health specialty workforce already in place in Mozambique.
  Interventions: Other: psychiatric medications and evidence-based psychotherapies
- Integrated Care (Experimental): Psychiatric medications and evidence-based psychotherapies to be provided by primary care providers.
  Interventions: Other: psychiatric medications and evidence-based psychotherapies
- Community Clinic Stepped Care (Experimental): Psychiatric medications and evidence-based psychotherapies to be provided by primary care providers and community health workers, respectively.
  Interventions: Other: psychiatric medications and evidence-based psychotherapies

INTERVENTIONS:
Other: psychiatric medications and evidence-based psychotherapies — Patients who screen positive with any psychiatric condition are referred for evaluation and treatment according to the treatment arm. This may combine psychiatric medications or evidence based psychotherapies according to treatment.

SUMMARY:
Global mental health (MH) and substance use disorders prevention, treatment and research gaps require that efficacious treatments be scaled-up, leveraging existing platforms. In tandem, participation of Ministries ready to apply evidence-inform policies must sustain them over time. PRIDE SSA may generate templates for other low- and middle-income countries (LMICs) by conducting a state of the art scale up study in Mozambique and by establishing a collaborative research network of nascent research "Seed Teams." Such "Seed Teams," trained by the capacity building component, may work across the region to build capacity and conduct implementation research to sustainably scale-up MH services. Scale Up Research (Mozambique) in MH and substance use disorders will evaluate strategies and costs of scaling up an innovative, integrated, sustainable, stepped-care community approach. The scale up study will leverage: (1) Mozambique's task-shifting strategy of training psychiatric technicians (PsyTs) to provide MH care, (2) the WHO-funded epilepsy community care program successfully implemented in 5 Provinces, now primed for scale-up by the Health Ministry. The cost-effective approach redefines work roles without requiring new human resources. Importantly, it comports with the Health Ministry's plan to implement prevention and treatment for all MH conditions, rather than single disorders. The model employs evidence-based practices (EBPs; e.g. Psychopharmacology; Interpersonal Therapy), already in use by PsyTs to: a) establish a sustainable program delivered and supervised by non-MH professionals, overseen by MH specialists; b) provide community screening, care and/or referrals for all MH disorders; and c) use implementation tools to monitor sustainability. This collaborative network will scale-up a cost-effective, sustainable program and inform policy.

DETAILED DESCRIPTION:
Working in three geographically separate Mozambican provinces and in rural (N=24), peri-urban (i.e., rural urban transition zone; N=6), and urban (N=6) clinics, the scale-up study first will conduct a two-year (12 months implementation, 12 months sustainability), cluster-randomized, three-arm hybrid effectiveness-implementation type 1 trial, guided by Proctor's implementation framework. The delivery pathway showing the highest overall effectiveness after this two-year trial in 36 clinics will then be implemented in clinics from the other two arms for two additional "cross-over" years. Throughout the trial and the "cross-over" years, qualitative and other process data will complement structured assessments to examine implementation, sustainability, and scale-up.

Scale-up PRIDES Mozambique has the following Specific Aims:

Aim 1. To determine the most effective delivery pathway in terms of 1) implementation outcomes (reach, retention, pathway fidelity, cost-effectiveness); 2) service-level outcomes (efficiency); and 3) patient-level outcomes (function/disability, comprehensive MH screener, patient satisfaction). As an Exploratory Sub-Aim: To assess the impact of: pre-implementation stage factors (acceptability, adoption); mediators (work self-efficacy, MH literacy); and moderators (clinic characteristics: rural, peri-urban, urban, epilepsy program implementation) on implementation, services, and patient outcomes.

Aim 2. To evaluate implementation, sustainability, and scale-up requirements of the most effective pathway (determined in Aim 1) in order to inform regional policies. A rigorous process evaluation mixed-methods approach will identify barriers and facilitators to implementing, sustaining, and scaling-up the most effective pathway in all clinics during the "cross-over" two years using purposive sampling for mixed-methods evaluation in a subset of 18 clinics (6 per Province).

Aim 3. To develop an implementation tool-kit for low-cost, feasible, and sustainable system-wide implementation of the most effective WHO Mental Health Gap Action Programme (mhGAP) delivery pathway in Sub-Saharan Africa (sSA) with collaboration of Members of the PRIDES sSA Five-Country Council, External Advisory Board and the WHO.

ELIGIBILITY:
Inclusion Criteria:

* Staff in one of the 36 clinics - Clinic directors, trainers, supervisors, providers of participating clinics: Community Health Workers; Nurses; and Medicine, Preventive Medicine andPsychiatric Technicians.

Exclusion Criteria:

* Other clinic staff besides clinic directors, trainers, supervisors, providers of participating clinics: Community Health Workers; Nurses; and Medicine, Preventive Medicine andPsychiatric Technicians.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Reach (implementation) | Change from Baseline in Reach at 12 months
  Number of people who access mental health care from those who need care
Cost | Cost of implementing each arm will be calculated through study completion, an average of 2 years
  Cost of Implementing each arm through the Stages of Implementation Completion (SIC) measure together with the Cost of Implementing New Strategies (COINS) method

SECONDARY OUTCOMES:
Change in Retention (implementation) | Change from Baseline in Retention at 12 months
  Number of people who receive mental health care from those who need care
Change in Clinical symptoms | Change from Baseline CmhTool at 12 months
  Symptom reduction using a newly validated tool - the Comprehensive Mental Health Tool (CmhTool) to monitor symptoms of common and severe mental disorders as well as substance use disorders

CONTACTS AND LOCATIONS:
Overall Officials: Milton L Wainberg, MD, Principal Investigator — NYSPI
Locations (1):
- MIHER: Mozambique Institute for Health Education and Research, Maputo, Cidade de Maputo, Mozambique

REFERENCES:
- [Background] Wainberg ML, Scorza P, Shultz JM, Helpman L, Mootz JJ, Johnson KA, Neria Y, Bradford JE, Oquendo MA, Arbuckle MR. Challenges and Opportunities in Global Mental Health: a Research-to-Practice Perspective. Curr Psychiatry Rep. 2017 May;19(5):28. doi: 10.1007/s11920-017-0780-z. PMID 28425023
- [Background] Dos Santos PF, Wainberg ML, Caldas-de-Almeida JM, Saraceno B, Mari Jde J. Overview of the mental health system in Mozambique: addressing the treatment gap with a task-shifting strategy in primary care. Int J Ment Health Syst. 2016 Jan 4;10:1. doi: 10.1186/s13033-015-0032-8. eCollection 2016. PMID 26734070
- [Derived] Wainberg ML, Lovero KL, Duarte CS, Fiks Salem A, Mello M, Bezuidenhout C, Mootz J, Feliciano P, Suleman A, Fortunato Dos Santos P, Weissman MM, Cournos F, Marques AH, Fumo W, Mabunda D, Alves-Bradford JE, Mello M, Mari JJ, Ngwepe P, Cidav Z, Mocumbi AO, Medina-Marino A, Wall M, Gouveia L, Oquendo MA. Partnerships in Research to Implement and Disseminate Sustainable and Scalable Evidence-Based Practices (PRIDE) in Mozambique. Psychiatr Serv. 2021 Jul 1;72(7):802-811. doi: 10.1176/appi.ps.202000090. Epub 2020 Dec 18. PMID 33334157